CLINICAL TRIAL: NCT02896361
Title: Burst Optimized Stimulation Study
Acronym: BOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Medizinische Einrichtungen der Universität Düsseldorf (Unknown); Klinikum Duisburg GmbH (Unknown); NKO Sint-Augustinus Antwerpen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJM-CIP-10125
Record Dates: First submitted 2016-09-01; First posted 2016-09-12 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stimulation order 1 (Experimental): Stimulations delivered in following order:
  1. Standard burst
  2. Burst Microdosing 1
  3. Burst Microdosing 2
  Interventions: Device: Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol
- Stimulation order 2 (Experimental): Stimulations delivered in following order:
  1. Burst Microdosing 1
  2. Burst Microdosing 2
  3. Standard burst
  Interventions: Device: Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol
- Stimulation order 3 (Experimental): Stimulations delivered in following order:
  1. Burst Microdosing 2
  2. Standard burst
  3. Burst Microdosing 1
  Interventions: Device: Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol

INTERVENTIONS:
Device: Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol — Stimulation parameters are reprogrammed from original values to study defined ones

SUMMARY:
This purpose of this study is to evaluate the therapeutic efficacy of burst microdosing stimulation paradigms in patients with chronic pain.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blinded crossover study designed to compare conventional burst stimulation parameters to two different burst microdosing paradigms.

Subjects will be randomized 1:1:1 to one of the three groups. Each group will evaluate all 3 stimulation paradigms in different order.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been implanted with a commercially available SJM spinal cord stimulator for controlling chronic intractable pain associated with back and/or leg pain;
* Subject has been exclusively using burst stimulation for at least three months;
* Subject is 18 years of age or older;
* Subject's pain-related medication regimen was stable in the 4 weeks prior to the screening evaluation;
* Subject agrees not to add or increase pain-related medication from enrollment through the study duration;
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all office visits;

Exclusion Criteria:

* Subject is currently participating in a clinical investigation study that includes an active treatment arm;
* Subject is currently receiving, applying or considering seeking workers compensation, or is involved in disability litigation;
* Subject has a non SJM neuromodulation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Venkatesan, Ph.D., Study Director — Abbott Medical Devices
Locations (3):
- NKO Sint-Augustinus, Antwerp, Belgium
- Germany (2):
  - Klinikum Duisburg GmbH, Duisburg, North Rhine-Westphalia
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 patients were screened for elegibility between july 2016 and may 2017 Dusseldorf (GER) and Wilrijk (BEL)
Pre-assignment Details: 27 of the 29 participants received the study intervention. Of those did not receive study intervention, 1 did not meet inclusion/exlusion criteria and 1 was withdrawn for non compliance.
Groups:
- Stimulation Order 1: Stimulations delivered in following order:
  1. Standard burst for 2 weeks
  2. Burst Microdosing 1 for 2 weeks
  3. Burst Microdosing 2 for 2 weeks
  Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol: Stimulation parameters are reprogrammed from original values to study defined ones
- Stimulation Order 2: Stimulations delivered in following order:
  1. Burst Microdosing 1 for 2 weeks
  2. Burst Microdosing 2 for 2 weeks
  3. Standard burst for 2 weeks
  Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol: Stimulation parameters are reprogrammed from original values to study defined ones
- Stimulation Order 3: Stimulations delivered in following order:
  1. Burst Microdosing 2 for 2 weeks
  2. Standard burst for 2 weeks
  3. Burst Microdosing 1 for 2 weeks
  Reprogramming of spinal cord stimulator (Proclaim or Prodigy SJM internal pulse generator) parameters according to study protocol: Stimulation parameters are reprogrammed from original values to study defined ones
Period: First Intervention (2 Weeks)
Arm/Group | Stimulation Order 1 | Stimulation Order 2 | Stimulation Order 3
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Stimulation Order 1 | Stimulation Order 2 | Stimulation Order 3
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | Stimulation Order 1 | Stimulation Order 2 | Stimulation Order 3
Started | 9 | 10 | 8
Completed | 8 | 9 | 8
Not Completed | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — emergenge of several new painful regions | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline information collected from the two patients that exited the study before receiving intervention was included in the basline analysis
Groups:
- All Subjects: Baseline characteristics for all subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 17
  Belgium | 12

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Pain
Description: Standard evaluation of pain intensity. Scale goes from 0 to 100 millimiters. 0 means no pain, 100 means strongest imaginable pain
Time Frame: assessed every 2 weeks after each intervention, for a total of 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Microdosing A(5:5): Microdosing A: five seconds of Burst SCS alternating with five seconds of no stimulation
- Microdosing B: 5:10: Microdosing B: five seconds of Burst SCS alternating with ten seconds of no stimulation
- Continuous: Continuously delivered burst SCS
Arm/Group | Microdosing A(5:5) | Microdosing B: 5:10 | Continuous
Number analyzed (Participants) | 25 | 25 | 25
units on a scale | 46.88 (23.5) | 48.60 (21.48) | 46.76 (21.88)

2. Secondary Outcome: EQ-5D
Description: European Quality of life questionnaire 5 dimensions. Range goes from 0 to 1. 0 represents low quality of life, 1 represents high quality of life
Time Frame: assessed every 2 weeks after each intervention, for a total of 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing A(5:5) | Microdosing B: 5:10 | Continuous
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 0.59 (0.2) | 0.62 (0.19) | 0.59 (0.21)

3. Secondary Outcome: Subject Preference
Description: questionnaire to identify preferred stimulation paradigm. multiple choice questionnaire. Possible answers were
  * first intervention
  * second intervention
  * third intervention
  * no preference
Time Frame: assessed 6 weeks after baseline at the last follow up visit
Measure: Count of Participants; unit: Participants
Groups:
- Stimulation Order 1: Stimulations delivered in following order:
  1. Standard burst for 2 weeks
  2. Burst Microdosing 1 for 2 weeks
  3. Burst Microdosing 2 for 2 weeks
- Stimulation Order 2: Stimulations delivered in following order:
  1. Burst Microdosing 1 for 2 weeks
  2. Burst Microdosing 2 for 2 weeks
  3. Standard burst for 2 weeks
- Stimulation Order 3: timulations delivered in following order:
  1. Burst Microdosing 2 for 2 weeks
  2. Standard burst for 2 weeks
  3. Burst Microdosing 1 for 2 weeks
Arm/Group | Stimulation Order 1 | Stimulation Order 2 | Stimulation Order 3
Number analyzed (Participants) | 8 | 9 | 8
Participants
  first intervention | 2 | 1 | 3
  second intervention | 1 | 5 | 3
  third intervention | 2 | 2 | 1
  no preference | 3 | 1 | 1

4. Secondary Outcome: Subject Satisfaction
Description: questionnaire on satisfaction with current therapy
Time Frame: assessed every 2 weeks after each intervention, for a total of 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Microdosing A(5:5) | Microdosing B: 5:10 | Continuous
Number analyzed (Participants) | 25 | 25 | 25
Participants
  Dissatisfied | 3 | 5 | 7
  Neither satisfied or dissatisfied | 12 | 8 | 8
  satisfied | 9 | 10 | 7
  very dissatisfied | 1 | 1 | 2
  very satisfied | 0 | 1 | 1

5. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: assessed over 6 weeks of study participation
Measure: Number; unit: percentage of patients with AE
Arm/Group | All Subjects
Number analyzed (Participants) | 27
percentage of patients with AE | 3.7

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Standard Burst: reporting "per intervention" adverse events experienced while standard continuous burst was delivered
- Burst Microdosing 1: reporting "per intervention" adverse events experienced while burst microdosing 1 was delivered
- Burst Microdosing 2: reporting "per intervention" adverse events experienced while burst microdosing 2 was delivered
Arm/Group | Standard Burst | Burst Microdosing 1 | Burst Microdosing 2
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Burst (N=26) | Burst Microdosing 1 (N=27) | Burst Microdosing 2 (N=26)
Bilateral ISG syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — One subject reported an adverse event 35 days after randomization to Group 2. The subject developed a new pain condition, bilateral ISG syndrome after enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT02896361/Prot_SAP_000.pdf